CLINICAL TRIAL: NCT02187328
Title: Effect of Grapefruit Juice and Exercise on Cortisol Levels
Brief Title: Effects of Fruit Juices on Hormone Metabolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benedictine University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Ben-0614a
Record Dates: First submitted 2014-07-02; First posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Cortisol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Grapefruit juice (Experimental): 12.5 OZ Grapefruit juice: Subject will ingest grapefruit juice 12.5 OZ twice on the day of their scheduled laboratory visit. Once in the morning and once in the afternoon prior to their evening visit
  Interventions: Other: Grapefruit juice
- Apple juice (Placebo Comparator): 10.5 OZ Apple juice: Subject will ingest apple juice 10.5 OZ twice on the day of their scheduled laboratory visit. Once in the morning and once in the afternoon 3 hours prior to their evening visit.
  Interventions: Other: Apple juice

INTERVENTIONS:
Other: Grapefruit juice — Volunteers participate in two visits at least 5 days apart. The day of their visit they ingest 12.5 oz of grapefruit juice in the morning and 12.5 oz of grapefruit juice ingested in the afternoon, 3h before reporting to the laboratory. The order of the visits is randomized, one visit volunteers ingest apple juice only, the other visit grapefruit juice only
  Arms: Grapefruit juice
Other: Apple juice — Volunteers participate in two visits at least 5 days apart. The day of their visit they ingest 12.5 oz of grapefruit juice or Apple juice ingested in the morning and 12.5 oz of grapefruit juice ingested in the afternoon, 3h before reporting to the laboratory. The order of the visits is randomized, one visit volunteers ingest apple juice only, the other visit grapefruit juice only
  Arms: Apple juice

SUMMARY:
The purpose of this study is to determine whether grapefruit juice alters the metabolism of cortisol following intense exercise.

ELIGIBILITY:
Inclusion Criteria:

* Young men and women, not taking medications known to alter glucocorticoid metabolism

Exclusion Criteria:

* Diabetes, uncontrolled hypertension, obesity, any medication known to interact with grapefruit juice

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Plasma cortisol change from baseline at 45 minutes | Baseline, 45 minutes
  Plasma cortisol levels will be collected at baseline and 45 minutes post-exercise for the Grapefruit visit intervention and for the Apple juice intervention. The interventions are acute ( 1 day), there is no follow up. The interventions are at least 1 week apart. For a given subject, the estimated time for study completion for the 2 treatments is 14 to 30 days.

SECONDARY OUTCOMES:
Change in plasma cortisol from 15 minutes to baseline | baseline, 15 minutes
  Plasma cortisol levels will be collected at baseline and 15 minutes post-exercise for the Grapefruit visit intervention and for the Apple juice intervention. The interventions are acute ( 1 day), there is no follow up. The interventions are at least 1 week apart. For a given subject, the estimated time for study completion for the 2 treatments is 14 to 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Del Corral, PhD-MD, Principal Investigator — Benedictine University
Locations (1):
- Benedictine University, Lisle, Illinois, United States